CLINICAL TRIAL: NCT07021118
Title: The Use of Brain Computed Tomography in the Management of the Patient With Mild TBI in the Emergency Department
Brief Title: Mild TBI in the Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: TCL
Record Dates: First submitted 2025-05-29; First posted 2025-06-13 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Emergency Departments
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elegible population: Adult patients presenting to the emergency department for mild head trauma (Glasgow Coma Scale 13-15). Patients with trauma-related loss of consciousness lasting more than 30 minutes and patients with post-traumatic amnesia lasting more than 24 hours were excluded.

SUMMARY:
Mild TBI is one of the main causes of admission to the Emergency Department (ED). Brain computed tomography (CT) is one of the most widely used diagnostic tools to assess the presence of intracranial lesions. However, in Western countries, 85-95% of CT scans performed in the ED for mild TBI are negative. It is therefore conceivable that a significant number of CTs could be avoided by a more careful use of this exam. On the other hand, excessive use of CT exposes patients to unnecessary radiation, increases healthcare costs and slows down the management of patients in the ED.

This study aims to analyze the variability in the use of CT in mild TBI in Italian EDs, validate the scores designed to help the physician decide when to use it and develop a model that predicts the medium-term outcome of patients with mild head trauma.

DETAILED DESCRIPTION:
Mild TBI is one of the most frequent causes of emergency department (ED) admission and is characterized by an increasing incidence. Brain computed tomography (CT) is a fundamental diagnostic tool to assess the presence and extent of any brain lesions and is commonly used in the ED for timely diagnosis. In particular, it allows to identify structural damage, such as hemorrhages, which could put the patient's life at risk if not treated promptly. However, the use of CT involves exposure to ionizing radiation, increases healthcare costs and can slow down the flow of patients in the ED. Considering that it is estimated that between 85% and 95% of patients with mild TBI do not have any brain lesions, a careful clinical evaluation is essential in indicating this investigation. These elements generate significant variability in the use of CT in mild TBI.

Several families of criteria and guidelines have been developed to support clinical decisions in this area, including the Canadian CT Head Rule, the Nexus II criteria, the New Orleans criteria and the National Institute for Health and Care Excellence (NICE) guidelines on head trauma. Although these criteria have been validated in multiple studies, their main objective is the identification of positive CT. This represents a limitation, since in many cases marginal brain injuries do not cause clinically relevant consequences or require specific interventions or treatments.

In this context, the present study aims to answer several research questions. First, the variability of CT use in Italian EDs will be analyzed, with the aim of identifying any discrepancies and the factors that determine them. The ultimate goal is to improve the quality of care for patients with mild head trauma. Second, the validity of the main tools proposed in the literature to support the clinical decision on the use of CT will be evaluated. Finally, the study aims to develop a new decision-making tool that can help ED physicians identify patients at risk of clinically relevant events in the short term, in order to facilitate a more accurate use of CT.

ELIGIBILITY:
Inclusion Criteria:

Adult patients arriving in the emergency department. Adult patients with mild TBI Adult patients with Glasgow Coma Scale 13-15.

Exclusion Criteria:

All patients under 18 years. Patients with trauma-associated loss of consciousness lasting more than 30 minutes.

Patients with post-traumatic amnesia lasting more than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients arriving in the emergency department with mild TBI (Glasgow Coma Scale 13-15). Patients with trauma-associated loss of consciousness lasting more than 30 minutes and patients with post-traumatic amnesia lasting more than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
To assess the use of CT | September 2025 - August 2026
  The heterogeneity of CT use between centers will be assessed using the Pearson chi-square test. If significant heterogeneity in the case-mix of patients between EDs emerges, this crude analysis will be supported by a standardized analysis. Specifically, the Standardized Event Ratio (SER) will be calculated for each ED, i.e. the ratio between CT performed in a center and those expected based on the characteristics of patients arriving at that ED. The number of expected CBTs will be calculated using a logistic regression model, developed on all patients enrolled in the study.

SECONDARY OUTCOMES:
Validate the most common scores | September 2026 - August 2027
  The scores will be evaluated primarily on the basis of sensitivity with respect to the positivity of patients to CT. In fact, since these scores are developed with the aim of identifying patients for whom CT may not be performed safely, it is essential that the scores identify as positive all patients who present a lesion to CT, or that have a very high sensitivity. Secondary indicators of performance of the scores will be the specificity and the ROC curve with respect to the positivity of CT, and sensitivity, specificity and ROC curve with respect to the presence of a clinically relevant outcome at 30 days. Subgroup analyses are planned to evaluate the performance of the scores on patients taking antiplatelet and/or anticoagulant therapies or with coagulation disorders.
Develop a new score to improve existing ones. | January 2027 - August 2027
  The development of a new score to guide the use of CT will be based on a multivariable logistic regression model. The outcome of interest will be the occurrence of clinically relevant events at 30 days from trauma in patients with positive CT. The variables collected in the study will be considered as candidate predictors and selected through a Least Absolute Shrinkage and Selection Operator (LASSO) model, which represents one of the most robust approaches to identify relevant predictors even in contexts where the number of candidate predictors is high compared to the sample size. The coefficients obtained from the model will be used to construct a composite score to estimate the probability of developing clinically relevant events at 30 days from mild head trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Milano Ospedale Maggiore, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided